CLINICAL TRIAL: NCT03358602
Title: Radiotherapy Versus Elective Neck Dissection for Management of Cervical Nodes in Clinical T1/2N0 Supraglottic Squamous Cell Carcinoma
Brief Title: Radiotherapy vs Neck Dissection for Clinical T1/2N0 Supraglottic Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Tianjin Medical University General Hospital (Other); Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJLC-01
Record Dates: First submitted 2017-11-21; First posted 2017-11-30 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Supraglottic Cancer
Keywords: Supraglottic cancer; Laryngeal cancer; Cervical lymph node; Neck dissection
MeSH Terms: conditions — Laryngeal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy (Experimental): Radiotherapy & open partial supraglottic laryngectomy(primary tumor)
  Interventions: Radiation: Radiotherapy
- Elective neck dissection (Active Comparator): Elective neck dissection & open partial supraglottic laryngectomy(primary tumor)
  Interventions: Procedure: Selective neck dissection

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy with a dose of 66-70 Gy is used to manage the cervical lymph nodes
  Arms: Radiotherapy
Procedure: Selective neck dissection — Selective neck dissection, defined as surgical clearance of the upper jugular (leveI II), midjugular (level III) and sometimes submandibular (level I) nodes, is used to manage the cervical lymph nodes
  Arms: Elective neck dissection

SUMMARY:
Supraglottic cancer is a main type of laryngeal carcinoma, which is one of the most common head and neck tumors. Cervical nodal metastasis is an important prognostic factor in supraglottic cancer. Current management, following the US National Comprehensive Cancer Network guidelines for T1-2, N0 supraglottic cancer (NCCN 2017), is either definitive radiotherapy or primary surgery with or without neck dissection. The optimal neck treatments strategy remains unclear in clinical settings owing to the limitation of a small number of retrospective studies and a lack of prospective trials. The investigators conducted a prospective, randomised trial to compare radiotherapy with neck dissection.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document
2. Age≥ 18 and≤ 75 years
3. Histological/ cytological/ Imaging examination proven supraglottic squamous-cell carcinoma in preoperative assessment
4. Cervical node negative according to the imaging characteristics and the physical examination
5. KPS≥ 70
6. Normal bone marrow reserve function and normal liver, kidney function
7. Expected survival period≥ 12 months

Exclusion Criteria:

1. Inability to provide an informed consent
2. Proved distant metastasis
3. Clinical stage 3-4
4. The patient has received prior surgery or radiotherapy (except for biopsy )
5. The patient has received chemotherapy(including targeted therapies) or immunotherapy
6. Prior malignancy within the previous 5 years
7. Severe mental disorders
8. Pregnant or lactating women
9. Other disease requiring simultaneous surgery or radiotherapy
10. Researchers believe that the situation is unsuitable for participation in the group

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2017-12-20 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Neck control rates | 2 years
  The percentage of patients without cervical lymph node metastasis

SECONDARY OUTCOMES:
Disease-free survival | 1 year
  The proportion of patients did not find clear evidence of recurrence or metastasis
Disease-free survival | 2 years
  The proportion of patients did not find clear evidence of recurrence or metastasis
Disease-free survival | 3 years
  The proportion of patients did not find clear evidence of recurrence or metastasis
Disease-free survival | 5 years
  The proportion of patients did not find clear evidence of recurrence or metastasis
Overall survival | 3 years
  The proportion of patients who survived
Overall survival | 5 years
  The proportion of patients who survived
Quality of life (EORTC QLQ-C30) | 1 year
  Evaluated by the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30
Quality of life (EORTC QLQ-HN35) | 1 year
  Evaluated by the European Organization for Research and Treatment of Cancer (EORTC) QLQ-HN35
Treatment cost | 4 weeks
  The total cost of the treatment of the primary and cervical lymph nodes until the discharge

CONTACTS AND LOCATIONS:
Overall Officials: Lun Zhang, Ph.D, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hopital, Tianjin, Tianjin Municipality, China